CLINICAL TRIAL: NCT01540136
Title: A Randomized Phase III Non-inferiority Study of Concurrent Chemoradiotherapy With Nedaplatin Versus Cisplatin in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Concurrent Chemoradiotherapy With Nedaplatin Versus Cisplatin in Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Medical University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Meizhou City Hospital Of Guangdong Provience (Unknown)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sun Yat-sen University
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2013-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nedaplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nedaplatin (Experimental): Nedplatin combine with IMRT
  Interventions: Drug: Nedaplatin
- Cisplatin (Active Comparator): Cisplatin combine with IMRT
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Nedaplatin — Nedaplatin 100mg/m2(3 weekly),D1,D22,D43 of RT
  Other Names: NDP
  Arms: Nedaplatin
Drug: Cisplatin — Cisplatin 100mg/m2(3 weekly),D1,D22,D43 of RT
  Other Names: DDP
  Arms: Cisplatin

SUMMARY:
This is a Phase III trial to study the effectiveness of nedaplatin versus cisplatin with IMRT chemoradiotherapy in treating patients with locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China and Southeast Asia. Several prospective randomized trials have demonstrated that concurrent chemoradiotherapy was superior to radiotherapy alone in the treatment of locoregionally advanced NPC. Cisplatin-based chemotherapy has been shown to have higher response rates in NPC than noncisplatin regimens. However, the patients' compliance was unsatisfactory because the obvious gastrointestinal toxicity of cisplatin. Nedaplatin is the new second generation platinum and it has slight gastrointestinal reaction. Our trial is in order to study the effectiveness of nedaplatin or cisplatin with intensity-modulated radiation therapy (IMRT) chemoradiotherapy in treating patients with locoregionally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Original clinical staged as T1-4N1-3 or T3-4N0（according to the 7th AJCC edition）
* No evidence of distant metastasis (M0)
* Male and no pregnant female
* Age between 18-65
* WBC ≥ 4,000/mm3 and PLT ≥ 100,000/mm3
* With normal liver function test (ALT、AST ≤ 2.5×ULN)
* With normal renal function test (Creatinine ≤ 1.5×ULN)
* Satisfactory performance status: Karnofsky scale (KPS)> 70
* Without radiotherapy or chemotherapy
* Patients must give signed informed consent

Exclusion Criteria:

* Patients have evidence of relapse or distant metastasis
* The presence of uncontrolled life-threatening illness
* Receiving other ways of anti-cancer therapy
* Receiving radiotherapy or chemotherapy
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Progress-free survival | 2 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site.

SECONDARY OUTCOMES:
Determine the toxic effects, both quantitatively and qualitatively, and quality of life (QoL) of these regimens in these patients. | 4 weeks
  Administration and Monitoring Patients will be evaluated in the clinic and eligibility and informed consent obtained. Patients will be monitored for clinical toxicity by standard NIH criteria. QoL was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) and EORTC QLQ Head and Neck. A time period of 4 weeks will constitute the time for clinical safety monitoring.
Complete Response (CR) | after the completion of the chemoradiotherapy treatment (up to 9 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the chemoradiotherapy treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only.
Overall Survival(OS) | 2 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival(LRRFS) | 2 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant Metastasis-Free Survival (DMFS) | 2 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Anti-neoplasms sensitization effects of chemotherapy to radiotherapy | radiotherapy in 20Gy、40Gy、70Gy
  Tumor response will be evaluated by physical examination and nasopharyngoscopy when radiotherapy in 20Gy、40Gy、70Gy.
Cost-effectiveness analysis | completion of chemoradiotherapy
  The determination of cost, including direct cost drug fees, inspection fees, expenses and nursing cost; cost-effectiveness analysis, such as cost-effectiveness ratio (ratio of the direct cost and short - and long-term curative effect) and incremental cost-effectiveness ratio (i.e., increasing costs and increase short or long-term efficacy ratio).
Correlate effects of CCRT with biomarkers of response and predictors of long-term outcome | before chemoradiotherapy and after chemoradiotherapy
  Early identification of patients who will have more aggressive disease soon after diagnosis has been a major goal, we will investigate the correlate effects of CCRT with biomarkers of response and predictors of long-term outcome in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: HaiQiang Mai, MD,Ph.D, Principal Investigator — Cancer center
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zheng J, Wang G, Yang GY, Wang D, Luo X, Chen C, Zhang Z, Li Q, Xu W, Li Z, Wang D. Induction chemotherapy with nedaplatin with 5-FU followed by intensity-modulated radiotherapy concurrent with chemotherapy for locoregionally advanced nasopharyngeal carcinoma. Jpn J Clin Oncol. 2010 May;40(5):425-31. doi: 10.1093/jjco/hyp183. Epub 2010 Jan 19. PMID 20085903
- [Background] Fuwa N, Kodaira T, Tachibana H, Nakamura T, Daimon T. Dose escalation study of nedaplatin with 5-fluorouracil in combination with alternating radiotherapy in patients with head and neck cancer. Jpn J Clin Oncol. 2007 Mar;37(3):161-7. doi: 10.1093/jjco/hyl138. Epub 2007 Mar 1. PMID 17332057
- [Background] Tanaka T, Yukawa K, Umesaki N. Radiation reduces carboplatin sensitivity and enhances nedaplatin sensitivity in cervical squamous cell carcinoma in vitro. Eur J Gynaecol Oncol. 2007;28(5):352-5. PMID 17966212
- [Background] Chen QY, Wen YF, Guo L, Liu H, Huang PY, Mo HY, Li NW, Xiang YQ, Luo DH, Qiu F, Sun R, Deng MQ, Chen MY, Hua YJ, Guo X, Cao KJ, Hong MH, Qian CN, Mai HQ. Concurrent chemoradiotherapy vs radiotherapy alone in stage II nasopharyngeal carcinoma: phase III randomized trial. J Natl Cancer Inst. 2011 Dec 7;103(23):1761-70. doi: 10.1093/jnci/djr432. Epub 2011 Nov 4. PMID 22056739
- [Background] Chan AT, Teo PM, Ngan RK, Leung TW, Lau WH, Zee B, Leung SF, Cheung FY, Yeo W, Yiu HH, Yu KH, Chiu KW, Chan DT, Mok T, Yuen KT, Mo F, Lai M, Kwan WH, Choi P, Johnson PJ. Concurrent chemotherapy-radiotherapy compared with radiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: progression-free survival analysis of a phase III randomized trial. J Clin Oncol. 2002 Apr 15;20(8):2038-44. doi: 10.1200/JCO.2002.08.149. PMID 11956263
- [Background] Ma J, Mai HQ, Hong MH, Min HQ, Mao ZD, Cui NJ, Lu TX, Mo HY. Results of a prospective randomized trial comparing neoadjuvant chemotherapy plus radiotherapy with radiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma. J Clin Oncol. 2001 Mar 1;19(5):1350-7. doi: 10.1200/JCO.2001.19.5.1350. PMID 11230478
- [Derived] Tang QN, Liu LT, Qi B, Guo SS, Luo DH, Sun R, Sun XS, Chen DP, Guo L, Mo HY, Wang P, Liu SL, Liang YJ, Li XY, Yang ZC, Chen QY, Mai HQ, Tang LQ. Effect of Concurrent Chemoradiotherapy With Nedaplatin vs Cisplatin on the Long-term Outcomes of Survival and Toxic Effects Among Patients With Stage II to IVB Nasopharyngeal Carcinoma: A 5-Year Follow-up Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2138470. doi: 10.1001/jamanetworkopen.2021.38470. PMID 34928359
- [Derived] Tang LQ, Chen DP, Guo L, Mo HY, Huang Y, Guo SS, Qi B, Tang QN, Wang P, Li XY, Li JB, Liu Q, Gao YH, Xie FY, Liu LT, Li Y, Liu SL, Xie HJ, Liang YJ, Sun XS, Yan JJ, Wu YS, Luo DH, Huang PY, Xiang YQ, Sun R, Chen MY, Lv X, Wang L, Xia WX, Zhao C, Cao KJ, Qian CN, Guo X, Hong MH, Nie ZQ, Chen QY, Mai HQ. Concurrent chemoradiotherapy with nedaplatin versus cisplatin in stage II-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2018 Apr;19(4):461-473. doi: 10.1016/S1470-2045(18)30104-9. Epub 2018 Feb 28. PMID 29501366
- See also: cancer — http://www.nlm.nih.gov/medlineplus/
- See also: cisplatin — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: nedaplatin — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp